CLINICAL TRIAL: NCT03423173
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Demonstrate Lot-to-Lot Consistency of 3 Lots of a Tetravalent Dengue Vaccine Candidate in Healthy Adults in Non-Endemic Country(Ies) for Dengue
Brief Title: Lot-to-lot Consistency of 3 Lots of Tetravalent Dengue Vaccine (TDV) in Non-endemic Country(Ies) for Dengue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEN-304
Record Dates: First submitted 2018-01-31; First posted 2018-02-06 (Actual); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Dengue Fever
Keywords: Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): TDV placebo matching injection, subcutaneously (SC) once on Day 1, and Day 90.
  Interventions: Biological: Placebo
- TDV Lot 1 (Experimental): Participants were administered TDV lot 1, 0.5 ml (each TDV 0.5 mL dose contained TDV-1, TDV-2, TDV-3, and TDV-4), SC injection, once on Day 1, and Day 90.
  Interventions: Biological: TAK-003
- TDV Lot 2 (Experimental): Participants were administered TDV lot 2, 0.5 ml (each TDV 0.5 mL dose contained TDV-1, TDV-2, TDV-3, and TDV-4), SC injection, once on Day 1, and Day 90.
  Interventions: Biological: TAK-003
- TDV Lot 3 (Experimental): Participants were administered TDV lot 3, 0.5 ml (each TDV 0.5 mL dose contained TDV-1, TDV-2, TDV-3, and TDV-4), SC injection once on Day 1, and Day 90.
  Interventions: Biological: TAK-003

INTERVENTIONS:
Biological: TAK-003 — TDV subcutaneous injection
  Other Names: TDV
  Arms: TDV Lot 1; TDV Lot 2; TDV Lot 3
Biological: Placebo — TDV Placebo-matching normal saline (0.9% NaCl) subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate lot-to-lot consistency in terms of equivalence of the immune responses induced by 3 consecutive TDV lots in healthy participants aged 18 to 60 years in non-endemic country(ies) for dengue.

DETAILED DESCRIPTION:
The vaccine tested in this study is Takeda's Tetravalent Dengue Vaccine Candidate (TDV). The primary objective of this trial is to investigate lot-to-lot consistency in terms of equivalence of the immune responses induced by 3 consecutive lots of TDV in healthy participants in non-endemic country(ies) for dengue.

The study will enroll approximately 924 healthy participants. Participants will be randomized in 2:2:2:1 to one of 4 trial groups to receive TDV (Lots 1, 2 or 3) or placebo:

* TDV 0.5 mL subcutaneous injection OR
* Placebo normal saline solution (0.9% NaCl) for injection.

In each trial group, all participants will receive 2 doses of TDV or placebo by subcutaneous injection on Days 1 (Month 0) and 90 (Month 3). Immunogenicity will be assessed in participants included in the immunogenicity subset (TDV groups: 176 participants each and placebo group: 88 participants) and safety will be assessed in all participants in each group.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is 270 days. Participants will make multiple visits to the clinic including a final visit at Day 270.

ELIGIBILITY:
Inclusion Criteria:

1. Is in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and the clinical judgment of the Investigator.
2. Signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.

Exclusion Criteria:

1. Has an elevated oral temperature (≥38°C or 100.4°F) within 3 days of the intended date of vaccination.
2. Known hypersensitivity or allergy to any of the vaccine components (including excipients of the investigational vaccine or placebo).
3. Has any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (e.g., Guillain-Barré syndrome).
4. Known or suspected impairment/alteration of immune function, including:

   1. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0) (use of inhaled, intranasal, or topical corticosteroids is allowed)
   2. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥ 2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0).
   3. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (M0) or planned administration during the trial.
   4. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
   5. Hepatitis C virus infection.
   6. Genetic immunodeficiency.
5. Has abnormalities of splenic or thymic function.
6. Has a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
7. Has any serious chronic or progressive disease according to judgment of the Investigator (e.g., neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
8. Has body mass index (BMI) greater than or equal to 35 kg/m^2 (= weight in kg/[height in meters^2]).
9. Has history of substance or alcohol abuse within the past 2 years.
10. Had previous and planned vaccination (during the trial conduct) against any flavivirus including dengue, yellow fever (YF), Japanese encephalitis (JE) viruses or tick-borne encephalitis.
11. Has a current or previous infection with a flavivirus such as dengue, Zika, YF, JE, West Nile (WN) fever, tick-borne encephalitis or Murray Valley encephalitis and participants with a history of prolonged (≥1 year) habitation in a dengue endemic area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 923 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (14):
- United States (14):
  - Optimal Research, Huntsville, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Advanced Clinical Research, Boise, Idaho
  - Optimal Research, Peoria, Illinois
  - Synexus Limited- Council Bluffs, Council Bluffs, Iowa
  - Heartland Research Associates LLC - Augusta, Augusta, Kansas
  - Heartland Research Associates LLC, Park City, Kansas
  - Optimal Research, Rockville, Maryland
  - Synexus Limited - Minneapolis, Edina, Minnesota
  - Synexus Limited - St. Louis, St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Synexus Limited - Columbus, Columbus, Ohio
  - Advanced Clinical Research, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Rauscher M, Youard Z, Faccin A, Patel SS, Pang H, Zent O. Pregnancy outcomes following unintentional exposure to TAK-003, a live-attenuated tetravalent dengue vaccine. Expert Rev Vaccines. 2025 Dec;24(1):221-229. doi: 10.1080/14760584.2025.2480297. Epub 2025 Mar 27. PMID 40099800
- [Derived] Tricou V, Winkle PJ, Tharenos LM, Rauscher M, Escudero I, Hoffman E, LeFevre I, Borkowski A, Wallace D. Consistency of immunogenicity in three consecutive lots of a tetravalent dengue vaccine candidate (TAK-003): A randomized placebo-controlled trial in US adults. Vaccine. 2023 Nov 13;41(47):6999-7006. doi: 10.1016/j.vaccine.2023.09.049. Epub 2023 Oct 24. PMID 37884415

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in the United States from 12 February 2018 to 14 January 2019.
Pre-assignment Details: Healthy participants were enrolled in 2:2:2:1 ratio into one of the four trial groups and received either Tetravalent Dengue Vaccine (TDV) lot 1, TDV Lot 2, TDV Lot 3 or Placebo for the investigation of lot to lot consistency of three consecutive lots.
Period: Overall Study
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Started | 132 | 263 | 264 | 264
Received at Least 1 Dose of the IP (Investigational Product (IP) includes TDV and placebo.) | 131 | 263 | 262 (1 participant of TDV Lot 2 received vaccine of Lot 1 and was included in TDV Lot 1 in Safety Set.) | 263
Completed | 113 | 228 | 237 | 234
Not Completed | 19 | 35 | 27 | 30
Not completed — Randomized but not vaccinated | 1 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 10 | 19 | 17 | 22
Not completed — Withdrawal of consent | 4 | 10 | 4 | 5
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 2 | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants irrespective of whether a dose of the trial vaccine (TDV or placebo) was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3 | Total
Number analyzed (Participants) | 132 | 263 | 264 | 264 | 923
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (11.70) | 40.8 (12.54) | 42.0 (11.71) | 40.9 (12.77) | 41.2 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 144 | 150 | 134 | 497
  Male | 63 | 119 | 114 | 130 | 426
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 16 | 25 | 20 | 70
  Not Hispanic or Latino | 120 | 247 | 239 | 244 | 850
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2 | 4
  Asian | 3 | 2 | 4 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1 | 2
  Black or African American | 23 | 55 | 56 | 44 | 178
  White | 104 | 200 | 202 | 208 | 714
  More than one race | 0 | 5 | 2 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for height at Baseline.
  cm
    number analyzed (Participants) | 132 | 263 | 263 | 264 | 922
    (all) | 171.7 (10.67) | 171.0 (9.68) | 171.6 (10.11) | 171.8 (9.86) | 171.5 (9.99)
Weight [Mean (Standard Deviation); unit: kg] — Population: Number analyzed is the number of participants with data available for weight at Baseline.
  kg
    number analyzed (Participants) | 131 | 263 | 262 | 263 | 919
    (all) | 82.37 (15.275) | 79.63 (15.203) | 81.31 (16.543) | 82.35 (15.928) | 81.28 (15.827)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight (kg)/Height (m^2). Population: Number analyzed is the number of participants with data available for BMI at Baseline.
  kg/m^2
    number analyzed (Participants) | 131 | 263 | 262 | 263 | 919
    (all) | 27.84 (3.825) | 27.17 (4.270) | 27.50 (4.464) | 27.84 (4.408) | 27.55 (4.309)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 120 in the Immunogenicity Subset
Description: GMTs of neutralizing antibodies for each of the 4 Dengue Serotypes was measured by microneutralization test 50% [MNT50]. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: 1 month post second dose (Day 120)
Population: Per protocol Set (PPS) included all DENV-naïve participants in immunogenicity subset who received at least 1 dose of trial vaccine, with data available for Baseline (Day 1) and at least 1 post-Baseline immunogenicity measurement and had no major protocol violations.Number of participants analyzed:participants with data available at given timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 60 | 120 | 129 | 118
titer
  DENV-1 | 5.3 [4.7 to 6.1] | 202.9 [155.9 to 264.1] | 293.8 [214.9 to 401.6] | 322.1 [238.1 to 435.9]
  DENV-2 | 6.3 [4.8 to 8.2] | 3090.3 [2494.8 to 3828.0] | 2386.0 [1913.0 to 2976.1] | 3574.1 [3087.8 to 4137.0]
  DENV-3 | 5.4 [4.6 to 6.3] | 149.5 [116.6 to 191.6] | 117.3 [92.7 to 148.4] | 122.8 [97.4 to 155.0]
  DENV-4 | 5.4 [4.7 to 6.2] | 116.3 [93.8 to 144.2] | 187.9 [154.4 to 228.6] | 115.8 [94.0 to 142.5]
Statistical Analysis 1: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-1; Test type: Equivalence — Equivalence between immune responses of 2 trial groups was established if the 95% CI of the corresponding geometric mean ratio was within pre-specified equivalence margins of 0.5 and 2.0; Geometric Mean Titer (GMT) Ratio = 0.69, 95% CI 2-sided [0.46 to 1.04] — Analysis of variance (ANOVA) model was used for analysis, including natural logarithms of titers as a response variable and trial group as a factor
Statistical Analysis 2: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.91, 95% CI 2-sided [0.60 to 1.38] — ANOVA model was used for analysis, including natural logarithms of titers as a response variable and trial group as a factor
Statistical Analysis 3: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-1; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.63, 95% CI 2-sided [0.41 to 0.96] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.30, 95% CI 2-sided [0.98 to 1.71] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.67, 95% CI 2-sided [0.51 to 0.88] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-2; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.86, 95% CI 2-sided [0.65 to 1.15] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.27, 95% CI 2-sided [0.91 to 1.78] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.95, 95% CI 2-sided [0.68 to 1.33] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-3; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.22, 95% CI 2-sided [0.87 to 1.71] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-4; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 0.62, 95% CI 2-sided [0.46 to 0.82] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-4; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.62, 95% CI 2-sided [1.22 to 2.17] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-4; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; GMT Ratio = 1.00, 95% CI 2-sided [0.75 to 1.35] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants Who Are Seropositive for Each of the 4 Dengue Serotypes at Days 120 and 270 in the Immunogenicity Subset
Description: Seropositivity was defined as a reciprocal neutralizing titer ≥ 10. The 4 dengue virus serotypes were DENV-1, DENV-2, DENV-3 and DENV-4.
Time Frame: 1 month post second dose (Day 120) and 6 months post second dose (Day 270)
Population: PPS included all DENV-naïve participants in the immunogenicity subset who received at least 1 dose of trial vaccine, with data available for Baseline (Day 1) and at least 1 post-Baseline immunogenicity measurement, and who had no major protocol violations. Number analyzed are participants with data available at the given timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 63 | 124 | 131 | 124
percentage of participants
  DENV-1, Day 120: number analyzed (Participants) | 60 | 120 | 129 | 118
  DENV-1, Day 120 | 1.7 [0.0 to 8.9] | 97.5 [92.9 to 99.5] | 96.9 [92.3 to 99.1] | 99.2 [95.4 to 100.0]
  DENV-2, Day 120: number analyzed (Participants) | 60 | 120 | 129 | 118
  DENV-2, Day 120 | 6.7 [1.8 to 16.2] | 99.2 [95.4 to 100.0] | 98.4 [94.5 to 99.8] | 100.0 [96.9 to 100.0]
  DENV-3, Day 120: number analyzed (Participants) | 60 | 120 | 129 | 118
  DENV-3, Day 120 | 1.7 [0.0 to 8.9] | 97.5 [92.9 to 99.5] | 94.6 [89.1 to 97.8] | 98.3 [94.0 to 99.8]
  DENV-4, Day 120: number analyzed (Participants) | 60 | 120 | 129 | 118
  DENV-4, Day 120 | 1.7 [0.0 to 8.9] | 97.5 [92.9 to 99.5] | 100.0 [97.2 to 100.0] | 97.5 [92.7 to 99.5]
  DENV-1, Day 270: number analyzed (Participants) | 59 | 111 | 123 | 119
  DENV-1, Day 270 | 3.4 [0.4 to 11.7] | 97.3 [92.3 to 99.4] | 89.4 [82.6 to 94.3] | 95.8 [90.5 to 98.6]
  DENV-2, Day 270: number analyzed (Participants) | 59 | 111 | 124 | 120
  DENV-2, Day 270 | 6.8 [1.9 to 16.5] | 100.0 [96.7 to 100.0] | 97.6 [93.1 to 99.5] | 99.2 [95.4 to 100.0]
  DENV-3, Day 270: number analyzed (Participants) | 59 | 111 | 124 | 120
  DENV-3, Day 270 | 0 [0.0 to 6.1] | 95.5 [89.8 to 98.5] | 88.7 [81.8 to 93.7] | 92.5 [86.2 to 96.5]
  DENV-4, Day 270: number analyzed (Participants) | 59 | 111 | 123 | 120
  DENV-4, Day 270 | 0 [0.0 to 6.1] | 92.8 [86.3 to 96.8] | 94.3 [88.6 to 97.7] | 91.7 [85.2 to 95.9]
Statistical Analysis 1: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-1 at Day 120; Test type: Other; Seropositivity Rates Difference = 0.60, 95% CI 2-sided [-4.99 to 6.06] — 95% CI for the differences in seropositivity rates between TDV lots were calculated using the Newcombe and Wilson method
Statistical Analysis 2: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-1 at Day 120; Test type: Other; Seropositivity Rate Difference = -1.65, 95% CI 2-sided [-6.90 to 3.19] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-1 at Day 120; Test type: Other; Seropositivity Rate Difference = -2.25, 95% CI 2-sided [-7.45 to 2.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-1 at Day 270; Test type: Other; Seropositivity Rate Difference = 7.87, 95% CI 2-sided [0.64 to 15.30] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-1 at Day 270; Test type: Other; Seropositivity Rate Difference = 1.50, 95% CI 2-sided [-4.67 to 7.65] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-1 at Day 270; Test type: Other; Seropositivity Rate Difference = -6.37, 95% CI 2-sided [-14.00 to 1.04] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-2 at Day 120; Test type: Other; Seropositivity Rate Difference = 0.72, 95% CI 2-sided [-3.87 to 5.29] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-2 at Day 120; Test type: Other; Seropositivity Rate Difference = -0.83, 95% CI 2-sided [-5.24 to 3.17] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-2 at Day 120; Test type: Other; Seropositivity Rate Difference = -1.55, 95% CI 2-sided [-6.05 to 2.58] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-2 at Day 270; Test type: Other; Seropositivity Rate Difference = 2.42, 95% CI 2-sided [-2.12 to 7.44] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-2 at Day 270; Test type: Other; Seropositivity Rate Difference = 0.83, 95% CI 2-sided [-3.41 to 5.24] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-2 at Day 270; Test type: Other; Seropositivity Rate Difference = -1.59, 95% CI 2-sided [-6.67 to 3.17] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-3 at Day 120; Test type: Other; Seropositivity Rate Difference = 2.93, 95% CI 2-sided [-3.07 to 9.06] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-3 at Day 120; Test type: Other; Seropositivity Rate Difference = -0.81, 95% CI 2-sided [-6.17 to 4.44] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-3 at Day 120; Test type: Other; Seropositivity Rate Difference = -3.73, 95% CI 2-sided [-9.74 to 2.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-3 at Day 270; Test type: Other; Seropositivity Rate Difference = 6.79, 95% CI 2-sided [-1.03 to 14.56] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-3 at Day 270; Test type: Other; Seropositivity Rate Difference = 3.00, 95% CI 2-sided [-4.28 to 10.23] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-3 at Day 270; Test type: Other; Seropositivity Rate Difference = -3.79, 95% CI 2-sided [-11.97 to 4.39] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-4 at Day 120; Test type: Other; Seropositivity Rate Difference = -2.50, 95% CI 2-sided [-7.68 to 1.55] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-4 at Day 120; Test type: Other; Seropositivity Rate Difference = 0.04, 95% CI 2-sided [-5.47 to 5.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-4 at Day 120; Test type: Other; Seropositivity Rate Difference = 2.54, 95% CI 2-sided [-1.52 to 7.81] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-4 at Day 270; Test type: Other; Seropositivity Rate Difference = -1.52, 95% CI 2-sided [-9.14 to 5.69] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-4 at Day 270; Test type: Other; Seropositivity Rate Difference = 1.13, 95% CI 2-sided [-6.90 to 8.95] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-4 at Day 270; Test type: Other; Seropositivity Rate Difference = 2.64, 95% CI 2-sided [-4.68 to 10.18] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: GMTs of Neutralizing Antibodies for Each of the 4 Dengue Serotypes at Day 270 in the Immunogenicity Subset
Description: as for outcome 1
Time Frame: 6 months post second dose (Day 270)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 63 | 124 | 131 | 124
titer
  DENV-1: number analyzed (Participants) | 59 | 111 | 123 | 119
  DENV-1 | 5.4 [4.9 to 5.9] | 122.5 [93.0 to 161.3] | 136.7 [95.2 to 196.3] | 168.4 [120.8 to 234.8]
  DENV-2: number analyzed (Participants) | 59 | 111 | 124 | 120
  DENV-2 | 5.8 [5.0 to 6.8] | 1507.2 [1242.3 to 1828.4] | 1097.5 [856.9 to 1405.5] | 1693.3 [1399.9 to 2048.3]
  DENV-3: number analyzed (Participants) | 59 | 111 | 124 | 120
  DENV-3 | NA [NA to NA] — Neutralizing antibodies were below the lower limit of detection (LLOD) and therefore geometric mean and 95% confidence interval couldn't be calculated. | 88.0 [69.2 to 111.9] | 63.1 [49.9 to 79.7] | 71.6 [57.3 to 89.5]
  DENV-4: number analyzed (Participants) | 59 | 111 | 123 | 120
  DENV-4 | NA [NA to NA] — Neutralizing antibodies were below the LLOD and therefore geometric mean and 95% confidence interval couldn't be calculated. | 64.1 [49.5 to 83.1] | 77.5 [60.8 to 98.8] | 51.2 [40.0 to 65.5]
Statistical Analysis 1: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-1; Test type: Other; GMT Ratio = 0.90, 95% CI 2-sided [0.56 to 1.42] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-1; Test type: Other; GMT Ratio = 0.81, 95% CI 2-sided [0.51 to 1.28] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-1; Test type: Other; GMT Ratio = 0.73, 95% CI 2-sided [0.46 to 1.16] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-2; Test type: Other; GMT Ratio = 1.37, 95% CI 2-sided [1.02 to 1.86] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-2; Test type: Other; GMT Ratio = 0.65, 95% CI 2-sided [0.48 to 0.87] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-2; Test type: Other; GMT ratio = 0.89, 95% CI 2-sided [0.66 to 1.21] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-3; Test type: Other; GMT Ratio = 1.40, 95% CI 2-sided [1.00 to 1.94] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-3; Test type: Other; GMT Ratio = 0.88, 95% CI 2-sided [0.64 to 1.21] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-3; Test type: Other; GMT Ratio = 1.23, 95% CI 2-sided [0.88 to 1.71] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: TDV Lot 1 vs TDV Lot 2; DENV-4; Test type: Other; GMT Ratio = 0.83, 95% CI 2-sided [0.58 to 1.18] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: TDV Lot 2 vs TDV Lot 3; DENV-4; Test type: Other; GMT Ratio = 1.51, 95% CI 2-sided [1.07 to 2.14] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: TDV Lot 1 vs TDV Lot 3; DENV-4; Test type: Other; GMT Ratio = 1.25, 95% CI 2-sided [0.88 to 1.78] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Percentage of Participants With Solicited Local (Injection Site) Adverse Events (AEs) by Severity After Each Vaccination
Description: Solicited local AEs (at injection site) were collected by participants using diary cards within 7 days after vaccination and included pain (none, mild: no interference with daily activity, moderate: interference with daily activity with or without treatment and severe: prevents daily activity with or without treatment), redness (erythema) (<25 mm, mild: >25 - ≤50 mm, moderate: >50 - ≤100 mm, severe: >100 mm) and swelling (edema/induration) (<25 mm, mild: >25 - ≤50 mm, moderate: >50 - ≤100 mm, severe: >100 mm ). The percentages were rounded off to the first decimal place.
Time Frame: Within 7 Days of each Vaccination (day of vaccination + 6 days)
Population: Safety Set included all participants who received at least 1 dose of trial vaccine (TDV or placebo). Participants were analyzed as treated. Number analyzed are participants with data available for the specific category. Only categories with at least one participant are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 131 | 264 | 261 | 263
percentage of participants
  After Vaccination 1, Any Local AE: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Any Local AE | 17.5 | 51.0 | 48.4 | 50.0
  After Vaccination 1, Pain-Any Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Pain-Any Severity | 16.7 | 45.5 | 40.6 | 41.7
  After Vaccination 1, Pain-Mild: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Pain-Mild | 15.0 | 39.9 | 34.8 | 37.7
  After Vaccination 1, Pain-Moderate: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Pain-Moderate | 1.7 | 5.5 | 5.1 | 4.0
  After Vaccination 1, Pain-Severe: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Pain-Severe | 0 | 0 | 0.8 | 0
  After Vaccination 1, Erythema-Any Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Erythema-Any Severity | 0.8 | 25.7 | 20.3 | 23.0
  After Vaccination 1, Erythema-Mild: 2.5-5(cm): number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Erythema-Mild: 2.5-5(cm) | 0 | 23.7 | 18.4 | 21.8
  After Vaccination 1,Erythema-Moderate: >5-<=10(cm): number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1,Erythema-Moderate: >5-<=10(cm) | 0 | 1.2 | 2.0 | 0.8
  After Vaccination 1, Erythema-Missing Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Erythema-Missing Severity | 0.8 | 0.8 | 0 | 0.4
  After Vaccination 1, Swelling-Any Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Swelling-Any Severity | 0.8 | 7.9 | 5.5 | 6.3
  After Vaccination 1, Swelling-Mild: 2.5-5(cm): number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Swelling-Mild: 2.5-5(cm) | 0 | 7.1 | 5.1 | 5.6
  After Vaccination 1,Swelling-Moderate: >5-<=10(cm): number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1,Swelling-Moderate: >5-<=10(cm) | 0 | 0.4 | 0.4 | 0
  After Vaccination 1, Swelling-Missing Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Swelling-Missing Severity | 0.8 | 0.4 | 0 | 0.8
  After Vaccination 2, Local AE-Any: number analyzed (Participants) | 115 | 232 | 240 | 237
  After Vaccination 2, Local AE-Any | 13.0 | 37.9 | 42.1 | 37.1
  After Vaccination 2, Pain-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Pain-Any Severity | 13.0 | 32.8 | 34.6 | 30.9
  After Vaccination 2, Pain-Mild: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Pain-Mild | 13.0 | 27.6 | 30.0 | 28.4
  After Vaccination 2, Pain-Moderate: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Pain-Moderate | 0 | 3.9 | 3.8 | 2.5
  After Vaccination 2, Pain-Severe: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Pain-Severe | 0 | 1.3 | 0.8 | 0
  After Vaccination 2, Erythema-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 237
  After Vaccination 2, Erythema-Any Severity | 0 | 19.0 | 18.8 | 14.3
  After Vaccination 2,Erythema-Mild: 2.5-5(cm): number analyzed (Participants) | 115 | 232 | 240 | 237
  After Vaccination 2,Erythema-Mild: 2.5-5(cm) | 0 | 18.1 | 17.1 | 13.1
  After Vaccination 2,Erythema-Moderate: >5-<=10(cm): number analyzed (Participants) | 115 | 232 | 240 | 237
  After Vaccination 2,Erythema-Moderate: >5-<=10(cm) | 0 | 0.4 | 1.7 | 1.3
  After Vaccination 2,Erythema-Missing Severity: number analyzed (Participants) | 115 | 232 | 240 | 237
  After Vaccination 2,Erythema-Missing Severity | 0 | 0.4 | 0 | 0
  After Vaccination 2, Swelling-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Swelling-Any Severity | 0 | 6.9 | 4.2 | 4.7
  After Vaccination 2,Swelling-Mild: 2.5-5(cm): number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2,Swelling-Mild: 2.5-5(cm) | 0 | 6.5 | 4.2 | 4.2
  After Vaccination 2,Swelling-Moderate: >5-<=10(cm): number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2,Swelling-Moderate: >5-<=10(cm) | 0 | 0 | 0 | 0.4
  After Vaccination 2,Swelling-Missing Severity: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2,Swelling-Missing Severity | 0 | 0.4 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Solicited Systemic Adverse Events (AEs) by Severity After Each Vaccination
Description: Solicited systemic AEs include fever, headache, asthenia, malaise and myalgia that occurred within 14 days after each vaccination. Solicited systemic AEs (headache, asthenia, malaise and myalgia) was graded from 0 to 3 by severity; where 0=None, 1=Mild: No interference with daily activity, 2=Moderate: Interference with daily activity, 3=Severe: Prevents daily activity; A systemic AE of fever (defined as ≥38°C or ≥100.4°F) was derived from a daily temperature reading recorded within 14 days after vaccination. Fever was excluded from the overall count as no severity grading was applied for it. The percentages were rounded off to the first decimal place.
Time Frame: Within 14 Days of each Vaccination (day of vaccination + 13 days)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 131 | 264 | 261 | 263
percentage of participants
  After Vaccination 1, Systemic AEs-Any: number analyzed (Participants) | 121 | 254 | 256 | 252
  After Vaccination 1, Systemic AEs-Any | 34.7 | 43.3 | 39.5 | 42.9
  After Vaccination 1, Headache-Any Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Headache-Any Severity | 22.5 | 28.9 | 27.0 | 28.6
  After Vaccination 1, Headache-Mild: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Headache-Mild | 17.5 | 21.3 | 19.9 | 21.4
  After Vaccination 1, Headache-Moderate: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Headache-Moderate | 4.2 | 5.9 | 5.5 | 6.0
  After Vaccination 1, Headache-Severe: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Headache-Severe | 0.8 | 1.6 | 1.6 | 1.2
  After Vaccination 1, Asthenia-Any Severity: number analyzed (Participants) | 120 | 252 | 256 | 252
  After Vaccination 1, Asthenia-Any Severity | 9.2 | 13.1 | 15.2 | 11.9
  After Vaccination 1, Asthenia-Mild: number analyzed (Participants) | 120 | 252 | 256 | 252
  After Vaccination 1, Asthenia-Mild | 7.5 | 7.9 | 9.4 | 6.3
  After Vaccination 1, Asthenia-Moderate: number analyzed (Participants) | 120 | 252 | 256 | 252
  After Vaccination 1, Asthenia-Moderate | 0.8 | 3.6 | 4.3 | 4.8
  After Vaccination 1, Asthenia-Severe: number analyzed (Participants) | 120 | 252 | 256 | 252
  After Vaccination 1, Asthenia-Severe | 0.8 | 1.6 | 1.6 | 0.8
  After Vaccination 1, Malaise-Any Severity: number analyzed (Participants) | 121 | 252 | 256 | 252
  After Vaccination 1, Malaise-Any Severity | 12.4 | 15.5 | 14.5 | 15.5
  After Vaccination 1, Malaise-Mild: number analyzed (Participants) | 121 | 252 | 256 | 252
  After Vaccination 1, Malaise-Mild | 9.1 | 7.1 | 7.8 | 8.3
  After Vaccination 1, Malaise-Moderate: number analyzed (Participants) | 121 | 252 | 256 | 252
  After Vaccination 1, Malaise-Moderate | 2.5 | 6.3 | 4.7 | 5.6
  After Vaccination 1, Malaise-Severe: number analyzed (Participants) | 121 | 252 | 256 | 252
  After Vaccination 1, Malaise-Severe | 0.8 | 2.0 | 2.0 | 1.6
  After Vaccination 1, Myalgia-Any Severity: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Myalgia-Any Severity | 15.8 | 26.5 | 25.4 | 22.2
  After Vaccination 1, Myalgia-Mild: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Myalgia-Mild | 13.3 | 19.0 | 16.0 | 14.3
  After Vaccination 1, Myalgia-Moderate: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Myalgia-Moderate | 2.5 | 7.1 | 7.8 | 7.5
  After Vaccination 1, Myalgia-Severe: number analyzed (Participants) | 120 | 253 | 256 | 252
  After Vaccination 1, Myalgia-Severe | 0 | 0.4 | 1.6 | 0.4
  After Vaccination 1, Fever-Any Severity: number analyzed (Participants) | 120 | 251 | 253 | 251
  After Vaccination 1, Fever-Any Severity | 1.7 | 0.8 | 2.4 | 2.0
  After Vaccination 1, Fever-38.0-<38.5: number analyzed (Participants) | 120 | 251 | 253 | 251
  After Vaccination 1, Fever-38.0-<38.5 | 0.8 | 0.4 | 0.8 | 1.2
  After Vaccination 1, Fever-38.5-<39.0: number analyzed (Participants) | 120 | 251 | 253 | 251
  After Vaccination 1, Fever-38.5-<39.0 | 0 | 0.4 | 0.8 | 0.8
  After Vaccination 1, Fever-39.0-<39.5: number analyzed (Participants) | 120 | 251 | 253 | 251
  After Vaccination 1, Fever-39.0-<39.5 | 0.8 | 0 | 0.4 | 0
  After Vaccination 1, Fever-≥41.0: number analyzed (Participants) | 120 | 251 | 253 | 251
  After Vaccination 1, Fever-≥41.0 | 0 | 0 | 0.4 | 0
  After Vaccination 2, Systemic AEs-Any: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Systemic AEs-Any | 23.5 | 26.7 | 29.2 | 28.0
  After Vaccination 2, Headache-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Headache-Any Severity | 19.1 | 18.1 | 22.5 | 18.6
  After Vaccination 2, Headache-Mild: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Headache-Mild | 15.7 | 15.1 | 15.8 | 13.6
  After Vaccination 2, Headache-Moderate: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Headache-Moderate | 3.5 | 3.0 | 5.4 | 4.2
  After Vaccination 2, Headache-Severe: number analyzed (Participants) | 115 | 232 | 240 | 236
  After Vaccination 2, Headache-Severe | 0 | 0 | 1.3 | 0.8
  After Vaccination 2, Asthenia-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Asthenia-Any Severity | 8.7 | 9.1 | 8.8 | 6.0
  After Vaccination 2, Asthenia-Mild: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Asthenia-Mild | 7.0 | 6.0 | 6.3 | 3.4
  After Vaccination 2, Asthenia-Moderate: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Asthenia-Moderate | 1.7 | 3.0 | 2.1 | 2.1
  After Vaccination 2, Asthenia-Severe: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Asthenia-Severe | 0 | 0 | 0.4 | 0.4
  After Vaccination 2, Malaise-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Malaise-Any Severity | 7.8 | 11.6 | 11.3 | 7.7
  After Vaccination 2, Malaise-Mild: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Malaise-Mild | 5.2 | 7.3 | 7.5 | 4.7
  After Vaccination 2, Malaise-Moderate: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Malaise-Moderate | 2.6 | 4.3 | 3.3 | 2.1
  After Vaccination 2, Malaise-Severe: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Malaise-Severe | 0 | 0 | 0.4 | 0.9
  After Vaccination 2, Myalgia-Any Severity: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Myalgia-Any Severity | 7.8 | 16.8 | 14.6 | 14.9
  After Vaccination 2, Myalgia-Mild: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Myalgia-Mild | 5.2 | 12.1 | 10.4 | 11.9
  After Vaccination 2, Myalgia-Moderate: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Myalgia-Moderate | 2.6 | 3.9 | 3.3 | 2.6
  After Vaccination 2, Myalgia-Severe: number analyzed (Participants) | 115 | 232 | 240 | 235
  After Vaccination 2, Myalgia-Severe | 0 | 0.9 | 0.8 | 0.4
  After Vaccination 2, Fever-Any Severity: number analyzed (Participants) | 115 | 231 | 240 | 234
  After Vaccination 2, Fever-Any Severity | 1.7 | 0.9 | 0.8 | 2.1
  After Vaccination 2, Fever-38.0-<38.5: number analyzed (Participants) | 115 | 231 | 240 | 234
  After Vaccination 2, Fever-38.0-<38.5 | 1.7 | 0.9 | 0.4 | 0.9
  After Vaccination 2, Fever-38.5-<39.0: number analyzed (Participants) | 115 | 231 | 240 | 234
  After Vaccination 2, Fever-38.5-<39.0 | 0 | 0 | 0.4 | 0.4
  After Vaccination 2, Fever-39.0-<39.5: number analyzed (Participants) | 115 | 231 | 240 | 234
  After Vaccination 2, Fever-39.0-<39.5 | 0 | 0 | 0 | 0.4
  After Vaccination 2, Fever-39.5-<40.0: number analyzed (Participants) | 115 | 231 | 240 | 234
  After Vaccination 2, Fever-39.5-<40.0 | 0 | 0 | 0 | 0.4

6. Secondary Outcome: Percentage of Participants With Any Unsolicited Adverse Events (AEs) After Each Vaccination
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.
Time Frame: Within 28 days (day of vaccination + 27 days) after each vaccination
Population: Safety Set included all participants who received at least 1 dose of trial vaccine (TDV or placebo). Participants were analyzed as treated. Number analyzed is the number of participants with data available for the specific category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 131 | 264 | 261 | 263
percentage of participants
  After First Vaccination | 13.7 | 18.6 | 18.0 | 16.7
  After Second Vaccination: number analyzed (Participants) | 116 | 237 | 247 | 243
  After Second Vaccination | 7.8 | 10.5 | 7.7 | 6.6

7. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, is an important medical event that may require intervention to prevent any of the above mentioned criteria and/or may expose the participant to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization. The percentages were rounded off to the first decimal place.
Time Frame: From the first vaccination on Day 1 until the end of the trial (Day 270)
Population: Safety Set included all participants who received at least 1 dose of trial vaccine (TDV or placebo). Participants were analyzed as treated.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 131 | 264 | 261 | 263
percentage of participants | 3.1 | 3.8 | 1.1 | 1.1

8. Secondary Outcome: Percentage of Participants With Medically Attended Adverse Events (MAAEs)
Description: MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional, including visits to an emergency department, but not fulfilling seriousness criteria. The percentages were rounded off to the first decimal place.
Time Frame: From the first vaccination on Day 1 until the end of the trial (Day 270)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
Number analyzed (Participants) | 131 | 264 | 261 | 263
percentage of participants | 13.7 | 17.8 | 12.3 | 11.8

ADVERSE EVENTS:
Time Frame: All-cause mortality and Serious adverse events: From the first vaccination on Day 1 until the end of the trial (Day 270); Other adverse events: Up to 28 days (Day of vaccination+27 subsequent days) after each vaccination.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Set included all participants who received at least 1 dose of trial vaccine (TDV or placebo). Participants were analyzed as treated.
Arm/Group | Placebo | TDV Lot 1 | TDV Lot 2 | TDV Lot 3
All-Cause Mortality (participants affected / at risk) | 1/131 | 0/264 | 0/261 | 0/263
Serious Adverse Events (participants affected / at risk) | 4/131 | 10/264 | 3/261 | 3/263
Other Adverse Events (participants affected / at risk) | 4/131 | 16/264 | 26/261 | 23/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | TDV Lot 1 (N=264) | TDV Lot 2 (N=261) | TDV Lot 3 (N=263)
Rhegmatogenous retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Anastomotic ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Perforation bile duct (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Infected seroma (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Chemical burn of gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 2 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=131) | TDV Lot 1 (N=264) | TDV Lot 2 (N=261) | TDV Lot 3 (N=263)
Injection site bruising (General disorders) | 1 | 5 | 10 | 12
Injection site pruritus (General disorders) | 0 | 8 | 15 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 6 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03423173/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT03423173/SAP_001.pdf